CLINICAL TRIAL: NCT01339780
Title: Imaging of Prostate and Breast Cancer Bone Metastases Using Magnetic Resonance Imaging and Nuclear Medicine Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Marko Seppanen, Dr., Turku University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 113/180/2010
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Bone Metastases
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- Breast Cancer (Experimental)
  Interventions: Radiation: BS, SPECT/CT, PET/CT, MRI
- Prostate Cancer (Experimental)
  Interventions: Radiation: BS, SPECT/CT, PET/CT, MRI

INTERVENTIONS:
Radiation: BS, SPECT/CT, PET/CT, MRI — Planar bone scintigraphy (BS), single photon emission computed tomography combined with low-dose computed tomography (SPECT/CT), 18F-fluoride positron emission tomography computed tomography (PET/CT) and magnetic resonance imaging (MRI) will be performed to all patients.

SUMMARY:
Prostate and breast cancer continues to be the most common cancer among men and women, respectively. The exact assessment of the cancer spread with detection of possible bone metastasis is crucial for treatment decision. In the current study 50 patients with prostate cancer and 50 patients with breast cancer at high risk for bone metastases or with know metastatic disease will be studied with multiple imaging modalities. Patients will be recruited from the Department of Oncology, Turku University Hospital. Planar bone scintigraphy (BS), single photon emission computed tomography combined with low-dose computed tomography (SPECT/CT), 18F-fluoride positron emission tomography computed tomography (PET/CT) and magnetic resonance imaging (MRI) will be performed to all patients. The primary objective is to determine the diagnostic accuracy of the four imaging modalities. The secondary goal is to calculate the sensitivities and specificities of the four imaging modalities on a patient-to-patient and lesion-to-lesion basis. Based on the results of this study an optimal imaging protocol for detection of prostate and breast cancer bone metastasis will be developed and validated.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 80 years
* Language spoken: Finnish or Swedish
* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* Diagnosis: Histologically confirmed prostate or breast cancer
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff
* strong suspicion of first bone metastatic disease (already diagnosed metastases in other organs, elevated tumor markers, destruction of bone in plain x-ray or otherwise specified reasons
* adjuvant chemo- or endocrine therapy is allowed

Exclusion Criteria:

* Ongoing treatment for metastatic disease
* Contraindications for MRI (cardiac pacemaker, intracranial clips etc.)
* Infections: Patient must not have an uncontrolled serious infection
* Claustrophobia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with bone metastases | at least 6 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Kiinamyllynkatu 4-8, Finland